CLINICAL TRIAL: NCT06527248
Title: Effects of Dietary Nitrate From Beetroot Juice on Vascular Function and Adaptations to Exercise Training in Postmenopausal Women: a Randomized, Placebo-controlled Study
Brief Title: Nitrate, Exercise and Vascular Function in Midlife Women
Acronym: Women's-Beet
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Collaborators: Medical University of Vienna (Other); Danube University Krems (Other); University of Giessen (Other); Edith Cowan University (Other); Flinders University (Other)
Responsible Party: Principal Investigator, Oliver Neubauer, Dr. (PhD) Priv.-Doz., University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UVienna_Women's-Beet
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Healthy; Menopause; Hypertension; Inflammation
Keywords: Women after menopause; Vascular function; Exercise training responsiveness; Cardiovascular health; Dietary nitrate-nitrite-nitric oxide-pathway; Beetroot juice
MeSH Terms: conditions — Hypertension; Inflammation

STUDY DESIGN:
Intervention Model Description: Prospective, mono-center, randomized, double-blind, placebo-controlled, parellel-group study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: One group will receive nitrate-rich beetroot juice and the other group will receive nitrate-depleted beetroot juice (as placebo) during the training period, on the background of a low-nitrate diet and an otherwise unaltered lifestyle. All products will be obtained from the same supplier (James White Drinks Ltd., UK). The nitrate-depleted beetroot juice is generated for research purposes only. The two juices will be indistinguishable by taste, color, smell and packaging. The investigators involved in the data acquisition and analysis will be blind to the trial allocation until the study has been completed and all analyses have been performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate group (Active Comparator): Daily consumption of 70 mL nitrate-rich beetroot juice concomitant with 12 weeks of exercise training
  Interventions: Dietary Supplement: Nitrate group
- Placebo group (Placebo Comparator): Daily consumption of 70 mL nitrate-depleted beetroot juice (placebo) concomitant with 12 weeks of exercise training
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Nitrate group — Daily consumption of 70 mL beetroot juice containing ~400 mg nitrate over an intervention period of 12 weeks concomitant to exercise training, either 3 hours pre-exercise on training days or with breakfast on non-training days.
  Other Names: Nitrate-rich beetroot juice
  Arms: Nitrate group
Dietary Supplement: Placebo group — Daily consumption of 70 mL nitrate-depleted beetroot juice (placebo) over an intervention period of 12 weeks concomitant to exercise training, either 3 hours pre-exercise on training days or with breakfast on non-training days.
  Other Names: Nitrate-depleted beetroot juice
  Arms: Placebo group

SUMMARY:
The purpose of this clinical study in women after menopause is to investigate whether the daily intake of nitrate from beetroot juice over 12 weeks enhances the positive effect of exercise training on vascular function, blood pressure and physical performance.

The risk of cardiovascular diseases (CVD) increases with advancing age and women are particularly affected. In women, the decline in the sex hormone oestrogen in the blood circulation with menopause contributes to impaired vascular function and an increased CVD risk; in part through increased inflammatory processes, oxidative stress, and a reduced body's own production of nitric oxide (NO). NO is a signaling molecule that is important for vascular function. Endurance-based exercise training is a key lifestyle strategy to prevent CVD. However, studies indicate that exercise is less effective in terms of its health-promoting adaptations in women after menopause as compared with men of similar age.

This study investigates the effect of exercise training in combination with the intake of nitrate-rich beetroot juice on functions of the cardiovascular system. Nitrate is a nitrogen compound that is found naturally in plant foods (e.g. beetroot juice) and is converted to NO in the human body. Results of previous studies indicate vasodilatory, blood pressure-lowering and performance-enhancing effects as well as positive influences on inflammatory processes and oxidative stress following nitrate intake. The hypothesis is that nitrate intake concomitant to training promotes training adaptations and further improves vascular function, blood pressure and physical performance compared to training without nitrate intake.

For the study, 54 untrained postmenopausal women (with the ages between 45 and 65 years) will be recruited and randomly allocated into two groups. Both groups will undergo 12 weeks of endurance-based exercise training. One group will receive nitrate-rich beetroot juice, and the other nitrate-depleted beetroot juice (as placebo). Vascular function, blood pressure, maximum oxygen uptake, and blood biomarkers for nitrate metabolism, inflammation status and oxidative stress will be examined.

The anticipated study results will provide new insights into whether nitrate as a 'training adjunct' improves health-promoting training adaptations in women after menopause. The overall aim is to improve the cardiovascular health and performance of middle-aged women and reduce their increased CVD risk.

DETAILED DESCRIPTION:
Wider research context:

Advancing age is a major risk factor for cardiovascular diseases (CVD). In women, the decline in the sex hormone oestrogen with menopause contributes to impaired vascular function and an increased CVD risk, in part via a reduced bioavailability of the endothelium-derived signaling molecule nitric oxide (NO), chronic low-grade inflammation and increased oxidative stress. Aerobic (or endurance) exercise training is a key lifestyle strategy to prevent CVD. However, data indicate that exercise is less effective for improving cardiovascular health in postmenopausal women as compared with men of similar age. Oestrogen treatment may restore vascular training adaptations but is associated with health risks. The main objective of this research is to examine whether dietary nitrate as a nutritional 'adjuvant' to regular exercise could be an innovative lifestyle intervention to favorably modulate vascular training adaptations and health in midlife women. This research expands upon findings by the investigators and others showing that inorganic nitrate from vegetables exerts benefits on physical function and cardiovascular health by increasing NO availability through the nitrate-nitrite-NO pathway and by attenuating inflammation and oxidative stress.

Objectives and hypotheses:

The investigators propose a clinical study to examine whether the daily consumption of nitrate-rich beetroot juice concomitant with aerobic exercise training improves vascular function, blood pressure, and cardiovascular fitness in postmenopausal women more effectively as compared with nitrate-depleted beetroot juice consumption (as placebo). The hypothesis is that the increased nitrate intake favorably modulates the systemic inflammatory and oxidative stress status and promotes cardiovascular health-related training outcomes.

Methods:

This study will involve a prospective, randomized, placebo-controlled parallel-group design. 54 untrained postmenopausal women (45-65 years) will be recruited and randomized into two groups. Both groups will undergo 12 weeks of endurance-based exercise training. The training will consist of a supervised training program that meets contemporary guidelines on aerobic physical activity. One group will receive nitrate-rich beetroot juice (containing ~400 mg nitrate, based on available evidence on the physiological and ergogenic benefits of nitrate), and the other nitrate-depleted beetroot juice (placebo), on the background of a low-nitrate diet and an otherwise unaltered lifestyle. 42 participants (21 per group) will be required to complete the study, based on power/sample size calculations with the forearm blood flow response to acetylcholine as primary endpoint. Secondary endpoints and additional measures will include 24 h-ambulatory blood pressure, maximal oxygen uptake, and blood inflammation and oxidative stress biomarkers.

Originality and innovation:

It is anticipated that this work will provide important new evidence on the efficacy of dietary nitrate to improve the training responsiveness, vascular function, and cardiovascular health in women after menopause. The objective of such a combined nutritional-training approach is to promote, preserve or restore physiological function and delay or possibly prevent the transition to functional limitations and CVD.

Research funding and cooperation arrangements:

This clinical research is funded by the Austrian Science Fund (FWF) (grant DOI 10.55776/KLP1075624). It is based on close collaborations between the University of Vienna and the Medical University of Vienna (both Austria), with the Department of Clinical Pharmacology at the Medical University of Vienna as the clinical trial center and Prof. M.D. Michael Wolzt as the coordinating physician of the trial center. The sponsor is the University of Vienna, as represented by the Principal Investigator Dr. Oliver Neubauer, Priv.-Doz. (Department of Nutritional Sciences, University of Vienna). Further national collaborations involve the groups of Prof. M.D. Daniel König, Prof. Karl-Heinz Wagner (both University of Vienna), and Prof. Viktoria Weber (University for Continuing Education Krems, Austria). International collaborations include Dr. Catherine P. Bondonno, Prof. Jonathan M. Hodgson (both Edith Cowan University), Prof. Richard J. Woodman (Flinders University) (all Australia), Prof. Karsten Krüger (Justus Liebig University of Giessen, Germany), and Prof. Jason D. Allen (University of Virginia, USA).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (amenorrhoeic ≥1 year), between the ages of 45 and 65 years, inclusive, who are either normotensive or are medically treated for stage 1 hypertension
* Written informed consent

Exclusion Criteria:

* Current or recent (within previous 3 months) engagement in exercise training (i.e., planned, structured, and regular exercise) with an average net exercise time of >2 hours per week
* Above-average cardiorespiratory fitness levels (i.e., a V̇O2 max max above the 75th percentile of age- and sex-specific normative data: ≥43 mL/kg/min for women aged 45-49 years, ≥38 mL/kg/min for women aged 50-59 years, ≥35 mL/kg/min for women aged 60-65 years)
* Any evidence of acute or chronic diseases such as symptomatic cardiovascular or peripheral vascular disease, moderate or severe chronic kidney disease (estimated glomerular filtration rate (GFR) <50 mL/min), pulmonary, neural, or musculoskeletal disease, osteoporotic fractures, cancer, or type 1 or 2 diabetes mellitus
* Fasting glucose >7.0 mmol/L or HbA1c > 6.5 rel. %
* BMI <18.5 kg/m2 or >30kg/m2
* A mean 24-hour ambulatory systolic/diastolic blood pressure of ≥130/80 mm Hg
* Irregular resting electrocardiography (ECG)
* Inability to perform physical exercise
* Abnormal cardiovascular responses during the baseline V ̇O2 max test, including symptoms, ECG abnormalities, arrhythmias, or exaggerated blood pressure responses
* Current or recent (<12 months) oestrogen-based hormone-replacement therapy
* Chronic use of nitric oxide (NO) donors, organic nitrites/nitrates, Ticagrelor, sodium-glucose cotransporter 2 (SGLT2) inhibitors, high-dose statins (i.e., Simvastatin >40mg/day, Atorvastatin >20mg/day, Rosuvastatin >10mg/day), acetylsalicylic acid >100mg/day, non-steroidal anti-inflammatory drugs (NSAID)
* A change in drug therapy likely to influence major outcomes within the previous 2 months, or likelihood that drug therapy would change during the study
* Use of antibiotics (within previous 2 months)
* Use of antibacterial mouthwash (volunteers willing to cease using antibacterial mouthwash for a period of 4 weeks before randomization will be included)
* Being vegan or vegetarian or consumption of >5 serves of vegetables per day
* Current or recent (within previous 6 months) significant (>6%) loss or gain of body weight
* Current or recent (<12 months) regular smoking of >5 cigarettes per day
* Alcohol intake of >70 g per week and/or binge drinking behaviour
* Inability or unwillingness to follow the study protocol

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Forearm blood flow (FBF) response to acetylcholine (FBFACh) | Change from baseline FBFACh to after the 12-week intervention period
  Endothelial-dependent microvascular function

SECONDARY OUTCOMES:
24-hour ambulatory systolic blood pressure | Change from baseline 24 hour-ambulatory systolic blood pressure to after the 12-week intervention period
  Ambulatory blood pressure monitoring
Maximal oxygen uptake (V̇O2 max) | Change from baseline V̇O2 max to after the 12-week intervention period
  Cardiorespiratory fitness: V̇O2 max

OTHER OUTCOMES:
FBF response to glyceryltrinitrate (FBFGTN) | Change from baseline FBFGTN to after the 12-week intervention period
  Endothelial-independent microvascular function
Clinic blood pressure | Change from baseline clinic blood pressure to after the 12-week intervention period
  Clinic blood pressure monitoring
Plasma and saliva nitrate and nitrite | Change from baseline plasma and saliva nitrate and nitrite to after the 12-week intervention period
  Nitrate metabolism: biomarker for nitrate bioavailability and functioning of the enterosalivary nitrate-nitrite-nitric oxide (NO) pathway
Serum hsCRP | Change from baseline hsCRP to after the 12-week intervention period
  Systemic inflammation status: serum high-sensitive C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Neubauer, Dr.Priv.Doz., Principal Investigator — University of Vienna

IPD SHARING:
Plan to Share IPD: Yes
For long-time preservation and sharing of the research data, it is planned to use the PHAIDRA digital repository of the University of Vienna (https://phaidra.univie.ac.at). This repository enables the permanent secure storage of digital assists including open access publications and research data necessary to reproduce and to verify the results of the publications.
  For all publications and other data related to this research that will be made available, all of the individual participant data collected during the trial will be de-identified.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The plan is to publish the findings in scientific journals and to present them at scientific meetings and to the public after the study is completed.
Access Criteria: Supporting the Open Access Policy of the University of Vienna, the PHAIDRA repository enables public access of the research data necessary to reproduce and to verify the results of publications from this research. The Austrian Science Fund (FWF) that funds this clinical research also requires to make peer-reviewed publications based on the results openly accessible on the Internet.

REFERENCES:
- [Background] Raubenheimer K, Bondonno C, Blekkenhorst L, Wagner KH, Peake JM, Neubauer O. Effects of dietary nitrate on inflammation and immune function, and implications for cardiovascular health. Nutr Rev. 2019 Aug 1;77(8):584-599. doi: 10.1093/nutrit/nuz025. PMID 31150091
- [Background] Woessner MN, McIlvenna LC, Ortiz de Zevallos J, Neil CJ, Allen JD. Dietary nitrate supplementation in cardiovascular health: an ergogenic aid or exercise therapeutic? Am J Physiol Heart Circ Physiol. 2018 Feb 1;314(2):H195-H212. doi: 10.1152/ajpheart.00414.2017. Epub 2017 Nov 3. PMID 29101174
- [Background] Shannon OM, Allen JD, Bescos R, Burke L, Clifford T, Easton C, Gonzalez JT, Jones AM, Jonvik KL, Larsen FJ, Peeling P, Piknova B, Siervo M, Vanhatalo A, McGawley K, Porcelli S. Dietary Inorganic Nitrate as an Ergogenic Aid: An Expert Consensus Derived via the Modified Delphi Technique. Sports Med. 2022 Oct;52(10):2537-2558. doi: 10.1007/s40279-022-01701-3. Epub 2022 May 23. PMID 35604567
- [Background] Moreau KL, Clayton ZS, DuBose LE, Rosenberry R, Seals DR. Effects of regular exercise on vascular function with aging: Does sex matter? Am J Physiol Heart Circ Physiol. 2024 Jan 1;326(1):H123-H137. doi: 10.1152/ajpheart.00392.2023. Epub 2023 Nov 3. PMID 37921669
- [Background] Baranauskas MN, Freemas JA, Tan R, Carter SJ. Moving beyond inclusion: Methodological considerations for the menstrual cycle and menopause in research evaluating effects of dietary nitrate on vascular function. Nitric Oxide. 2022 Jan 1;118:39-48. doi: 10.1016/j.niox.2021.11.001. Epub 2021 Nov 11. PMID 34774755
- [Background] Hogwood AC, Ortiz de Zevallos J, Weeldreyer N, Clark JR, Mazzella V, Cain L, Myaing D, Love KM, Weltman A, Allen JD. The acute effects of exercise intensity and inorganic nitrate supplementation on vascular health in females after menopause. J Appl Physiol (1985). 2023 Nov 1;135(5):1070-1081. doi: 10.1152/japplphysiol.00559.2023. Epub 2023 Oct 5. PMID 37795531
- [Background] Fejes R, Pilat N, Lutnik M, Weisshaar S, Weijler AM, Kruger K, Draxler A, Bragagna L, Peake JM, Woodman RJ, Croft KD, Bondonno CP, Hodgson JM, Wagner KH, Wolzt M, Neubauer O. Effects of increased nitrate intake from beetroot juice on blood markers of oxidative stress and inflammation in older adults with hypertension. Free Radic Biol Med. 2024 Sep;222:519-530. doi: 10.1016/j.freeradbiomed.2024.07.004. Epub 2024 Jul 5. PMID 38972612